CLINICAL TRIAL: NCT01366625
Title: Effects of Renal Denervation on Blood Pressure and Clinical Course of Obstructive Sleep Apnea in Patients With Resistant Hypertension
Brief Title: Renal Denervation in Patients With Resistant Hypertension and Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSA-Denerv1
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Hypertension; Obstructive Sleep Apnea
Keywords: hypertension, resistant; obstructive sleep apnea; renal denervation; continuous positive airway pressure therapy
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renal Denervation (Experimental): Renal Denervation and maintenance of anti-hypertensive medications and continuous positive airway pressure therapy
  Interventions: Device: Renal denervation with a catheter-based procedure (Symplicity® Catheter System)
- Maintenance of Medications (No Intervention): Maintenance of anti-hypertensive medications and continuous positive airway pressure therapy

INTERVENTIONS:
Device: Renal denervation with a catheter-based procedure (Symplicity® Catheter System) — Disruption of the renal nerves with a catheter-based procedure.
  Other Names: Renal Denervation (Symplicity® Catheter System)
  Arms: Renal Denervation

SUMMARY:
The purpose of this study is to investigate the clinical utility of renal denervation for the treatment of resistant hypertension coexisting with obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 and =< 70 years of age.
* systolic blood pressure >=140mmHg (office);
* on 3 or more antihypertensive medications (including diuretic)
* mean daytime systolic ABPM >= 135 mmHg
* obstructive sleep apnea (AHI >=15 event/hour, indications for CPAP treatment)

Exclusion Criteria:

* renal artery abnormalities
* eGFR < 60mL/min
* previous TIA, stroke, heart failure
* Type 1 diabetes
* ICD or pacemaker
* others

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2016-02-08 (Actual); Study Completion 2016-11-28 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Reduction | 3 months

SECONDARY OUTCOMES:
Responses to renal denervation (e.g., blood pressure reduction, sleep apnea course, metabolic assessment, cardiac changes) | Through 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Aleksander Prejbisz, M.D., Ph.D., Principal Investigator — Institute of Cardiology
Locations (1):
- Institute of Cardiology, Warsaw, Poland

REFERENCES:
- [Derived] Warchol-Celinska E, Prejbisz A, Kadziela J, Florczak E, Januszewicz M, Michalowska I, Dobrowolski P, Kabat M, Sliwinski P, Klisiewicz A, Topor-Madry R, Narkiewicz K, Somers VK, Sobotka PA, Witkowski A, Januszewicz A. Renal Denervation in Resistant Hypertension and Obstructive Sleep Apnea: Randomized Proof-of-Concept Phase II Trial. Hypertension. 2018 Aug;72(2):381-390. doi: 10.1161/HYPERTENSIONAHA.118.11180. Epub 2018 Jun 25. PMID 29941516